CLINICAL TRIAL: NCT03492905
Title: Implementation of Internet-based Cognitive Behaviour Therapy for Adolescents With Co-morbid Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Collaborators: Uppsala University (Other); Karolinska University (Other)
Responsible Party: Principal Investigator, Vendela Zetterqvist, licensed clinical psychologist, PhD, Uppsala University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2017/373
Record Dates: First submitted 2018-03-02; First posted 2018-04-10 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Masking Description: Outcome assessment is automatic, pre-programmed, on-line
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Internet-based CBT (Experimental): Internet-based Cognitive Behaviour Therapy (iCBT)
  Interventions: Behavioral: Internet-based Cognitive Behaviour Therapy (iCBT)

INTERVENTIONS:
Behavioral: Internet-based Cognitive Behaviour Therapy (iCBT) — Guided self-help for 7 weeks. Contact with therapist 2 times per week.

SUMMARY:
Insomnia is a commonly reported comorbidity for adolescents with psychiatric conditions. It is well-known that insomnia can exacerbate the concurrent psychiatric symptom load. Results from a pilot study shows that outpatients of Children and Youth Psychiatry can improve their sleep and depressive symptoms by receiving internet-based cognitive behavioral therapy for insomnia (iCBT). This study is designed to evaluate implementation of the treatment in routine care.The study will evaluate aspects of the implementation process such as organizational attitudes towards iCBT before implementation, level of knowledge about the condition and intervention among health-care providers before and after the implementation, and clinical outcomes in routine care.

ELIGIBILITY:
Inclusion Criteria:

* To fulfill the diagnostic criteria for insomnia
* To have access to a computer with Internet connection
* No previous or ongoing CBT for insomnia

Exclusion Criteria:

* Ongoing manic or psychotic episode
* Being at high risk of triggering manic or psychotic episode
* Ongoing sleep apnea

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI; Morin, 1993) | Pre-treatment, weekly for seven weeks (during treatment), after 7 weeks (i.e. post-treatment), after 7 weeks and 4 months (i.e. 4 months after treatment is completed)
  Change in severity of insomnia is assessed by measuring ISI at several measurement points before, during and after treatment. The score ranges from 0-28, higher values indicate worse symptoms of insomnia.

SECONDARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale - Self report (MADRS-S; Svanborg & Åsberg, 1994) | Pre-treatment, after 7 weeks (i.e. post-treatment), after 7 weeks and 4 months (i.e. 4 months after treatment is completed)
  Change in depressive symptoms is assessed by measuring MADRS-S at several measurement points before, during and after treatment. The score ranges from 0-35, higher values indicate worse symptoms of depression.
Childrens Global Assessment Scale (C-GAS; Shaffer et al., 1983) | Pre-treatment, after 7 weeks (i.e. post-treatment), after 7 weeks and 4 months (i.e. 4 months after treatment is completed)
  Change in clinician-rated level of functioning is assessed by measuring C-GAS at several measurement points before, during and after treatment. The score ranges from 0-100, higher values indicate better functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Vendela Zetterqvist, Ph D, Principal Investigator — Uppsala University Hospital
Locations (1):
- Uppsala University Hospital, Uppsala, Uppsala County, Sweden

IPD SHARING:
Plan to Share IPD: No